CLINICAL TRIAL: NCT04829903
Title: Dulaglutide Versus Liraglutide in Obese Type 2 Diabetic Adolescents Using Metformin: Results From a Randomized Double Blinded Clinical Trial
Brief Title: Dulaglutide Versus Liraglutide in Obese Type 2 Diabetic Adolescents Using Metformin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Dr Zainab Khan, Chief Resident, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DULACAI37628
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes Treated With Insulin; Obesity; Adolescent Obesity
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — dulaglutide; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group DUL (Active Comparator): Group taking Dulaglutide injections
  Interventions: Drug: Dulaglutide
- Group LIR (Placebo Comparator): Group taking Liraglutide injections
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Dulaglutide — Dulaglutide injections
  Other Names: Group DUL
  Arms: Group DUL
Drug: Liraglutide — Liraglutide injections
  Other Names: Group LIR
  Arms: Group LIR

SUMMARY:
To compare the efficacy and effect on glycemic control of Dulaglutide versus Liraglutide in obese Type 2 diabetic adolescents using metformin

DETAILED DESCRIPTION:
To observe the efficacy, effect on glycemic control, impact on BMI and incidence of adverse effects of Dulaglutide and to compare it to Liraglutide in individuals aged thirteen to eighteen who have Type 2 diabetes mellitus and are obese.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Obese
* Taking metformin
* Male or female

Exclusion Criteria:

* Non obese
* Not taking metformin
* Taking other injectable diabetic medications

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Glycemic level | 24 weeks for the duration of the study
  HbA1c
BMI | 24 weeks for the duration of the study
  BMI measurements using weight and height measurements (anthropometric)
Adverse effects | 24 weeks for the duration of the study
  Recording of adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Hussain, PhD, Principal Investigator — Al Ain University
Locations (1):
- Zainab Khan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No